CLINICAL TRIAL: NCT06241898
Title: A Phase I, Open Label, Multicenter, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of BB-1709 in Patients With Locally Advanced/Metastatic Solid Tumors
Brief Title: A First-in-human of Multiplle Doses of BB-1709 in Subjects With Locally Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bliss Biopharmaceutical (Hangzhou) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bliss
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dose escalation (Experimental): BB-1709 will be administered as an intravenous infusion by Q3W or Q2W as long as they continue to show clinical benefit as judged by the investigator, until disease progression or intolerable toxicity, withdrawal of consent, death, or termination of the study.
  Interventions: Drug: BB-1709
- dose expansion (Experimental): BB-1709 will be administered as an intravenous infusion by Q3W or Q2W as long as they continue to show clinical benefit as judged by the investigator, until disease progression or intolerable toxicity, withdrawal of consent, death, or termination of the study.
  Interventions: Drug: BB-1709

INTERVENTIONS:
Drug: BB-1709 — Subjects participating in Phase Ia study may continue to receive study treatment as long as they continue to show clinical benefit as judged by the investigator, until disease progression or intolerable toxicity, withdrawal of consent, death, or termination of the study.

SUMMARY:
The goal of this clinical trial is to test in patients with local advanced/metastatic solid tumors. the main questions it aims to answer are:

* to assess the safety and tolerability of BB-1709.
* to determine the maximum tolerated dose(MTD) and/or the PR2D of BB-1709

DETAILED DESCRIPTION:
The study consists of two parts: dose-escalation (Phase Ia) and dose expansion (Phase Ib).

Phase Ia is a multicenter, open-label, first time in human clinical trial to assess safety, tolerability, pharmacokinetics, immunogenicity, the preliminary anti-tumor activity of BB-1709, and to establish the MTD and/or RP2D of BB-1709 in patients with advanced solid tumors.

Phase Ib is to explore one or more RP2Ds to further assess safety, tolerability, pharmacokinetics, immunogenicity, and preliminary anti-tumor activity of BB-1709 in patients with specific types of solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent form (ICF) for the trial. Adult patients ≥ 18 years at the time of signing ICF.
2. Histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors in patients who must have progressed on, be refractory to, or intolerant to prior SOC.
3. At least one measurable lesion as defined per RECIST Version 1.1.
4. Be able to provide archived or fresh tumor tissue specimens.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy ≥12 weeks.

Exclusion Criteria:

1. Receiving anti-tumor therapy (systemic anti-tumor therapies, immunotherapy, biotherapy, topic therapy, other investigational product, radiation therapy, or surgery) within 4 weeks prior to the first dose of study treatment; receiving anti-tumor small-molecule agents within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of study treatment; receiving anti-tumor Chinese traditional medication and herbal remedies within 2 weeks prior to the first dose of study treatment.
2. Prior history of other malignancies within the previous 3 years, except for noninvasive malignancies such as cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, ductal carcinoma in situ of the breast that has been surgically cured.
3. Major surgery or significant traumatic injury within 4 weeks before the first dose of study treatment or not fully recovered from surgery; or surgery planned during the study.
4. Not recovered to baseline or CTCAE v5.0 ≤ grade 1 AEs from prior anti-cancer therapy except for alopecia, or asymptomatic and clinically not significant laboratory abnormalities.
5. Grade 2 or greater peripheral neuropathy (PN) when signing ICF, or history of grade 3 neurotoxicity or PN, or history of treatment discontinuation due to neurotoxicity or PN.
6. Active pneumonitis/interstitial lung disease (ILD), or history of radiotherapy to lung field within 12 months before the first dose of study treatment, or current lung disease with clinical symptoms(e.g., symptomatic chronic obstructive pulmonary disease or dyspnea)
7. Symptomatic or untreated central nervous system (CNS) metastases, or CNS metastases or leptomeningeal disease or carcinomatous meningitis requiring ongoing treatment for CNS metastases, including surgery or radiation therapy or steroids (>10 mg/day of prednisone or equivalent) and antiepileptic agents.
8. Uncontrolled ascites, pleural effusion or pericardial effusion, as determined by the Investigator.
9. Active autoimmune disease, except vitiligo or cured childhood asthma/allergies that requires no intervention after adulthood, autoimmune-mediated hypothyroidism treated with stable doses of thyroid hormone replacement, or Type I diabetes treated with stable doses of insulin can be excepted.
10. History of organ transplantation (i.e., stem cell or solid organ transplant).
11. Known history of human immunodeficiency virus (HIV) infection with the exception of patients with CD4+ T cell (CD4+) counts ≥350 cells/µL, or have not had a history of AIDS-defining opportunistic infections, or have not had a history of AIDS-defining opportunistic infections within the past 12 months , or on established antiretroviral therapy (ART) for more than four weeks and have an HIV viral load <400 copies/mL prior to enrollment.
12. Active hepatitis B or hepatitis C infection, demonstrated by positive serology or requiring treatment. Subjects who are anti-HBs/HBcAb (+) without detectable HBV-DNA or are with undetectable HCV RNA are eligible. Subjects co-infected with hepatitis B and hepatitis C should be excluded.
13. Any other serious underlying medical conditions, including but not limited to, uncontrolled diabetes mellitus, active uncontrolled infection (e.g. tuberculosis), active gastric ulcer, uncontrolled seizures, cerebrovascular incidents within 6 months prior to study treatment, gastrointestinal bleeding within 3 months prior to study treatment, severe signs and symptoms of coagulation and clotting disorders.
14. Receipt of live vaccines within 4 weeks prior to the first dose of the study drug.
15. Females who are pregnant or breastfeeding.
16. History of severe hypersensitivity or known to be allergic to protein drugs or recombinant proteins or excipients in BB-1709 drug formulation.
17. Concurrent condition that in the investigator's opinion would interfere with evaluation of the study drug or interpretation of subject safety or study results.

    -

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events | up to 3 years
  To evaluate the safety and tolerability of BB-1709

SECONDARY OUTCOMES:
Area under the serum concentration time curve from time 0 extrapolated to infinity (AUC0-inf) | Pre-dose and post-dose during Cycle 1 through Cycle 8. Duration of each cycle is 21 days
  To characterize the PK of BB-1709

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided